CLINICAL TRIAL: NCT01330719
Title: Mechanisms and Treatment Response of Aggressive Periodontitis in Children: Aberrant Immunological Phenotypes/Functions in the Progression of AgP
Brief Title: Mechanisms and Treatment Response of Aggressive Periodontitis in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB201400349-N; R01DE019456 (NIH)
Record Dates: First submitted 2011-04-04; First posted 2011-04-07 (Estimated); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Aggressive Periodontitis
Keywords: Periodontitis
MeSH Terms: conditions — Aggressive Periodontitis; Periodontitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diseased periodontal treatment (Experimental): Scaling and root planing along with systemic antibiotics (Amoxicillin 500 mg and Metronidazole 250 mg tid 7 days).
  Interventions: Procedure: Diseased periodontal treatment
- Conventional periodontal treatment (Active Comparator): Standard periodontal prophylaxis
  Interventions: Procedure: Conventional periodontal treatment

INTERVENTIONS:
Procedure: Diseased periodontal treatment — Treatment includes scaling and root planing with systemic antibiotics, Amoxicillin 500 mg and Metronidazole 250 mg tid 7 days. At certain intervals after the scaling and root planing, your gums will be reevaluated. You will receive further surgical gum therapy only if your gums haven't shown improvement after first treatment on the reevaluation appointments. If surgery is needed, a bone substituting material may be necessary to "fill" the spaces where bone has been destroyed by the disease. Extraction of teeth might also be part of gum treatment if the disease is very severe. Re-treatment with antibiotics also may be necessary depending on the response after treatment. You are usually re-examined and receive additional cleanings every 3 to 6 months to ensure the disease does not come back.
  Arms: Diseased periodontal treatment
Procedure: Conventional periodontal treatment — Scaling and gum measurement will be taken to compare to the treated group.- If it is determined that you do not have this disease, a conventional cleaning is done, usually every 6 months. This is all part of normal clinical care.
  Arms: Conventional periodontal treatment

SUMMARY:
Although of low prevalence, aggressive periodontitis is a rapid destructive form of periodontal disease that initiates at a young age, leading to premature loss of first molars and incisors. Little is known on the mechanisms of this disease. It is imperative to understand mechanisms of disease to establish proper treatment. We have established a controlled study in a comparable population presenting similar aggressive disease characteristics to evaluate the mechanisms of this disease. It is the goal of this study to determine immunological and microbiological mechanisms responsible for the rapid tissue destruction in children with localized aggressive periodontitis and how traditional periodontal intervention affects these mechanisms. Important knowledge gained with this proposal will aid in defining specific treatment approaches to better control disease progression and prevent disease initiation in susceptible individuals.

DETAILED DESCRIPTION:
There a multiple appointments throughout the study which can vary depending upon if a patient has the disease present or not.

If the patient has gum disease: At the initial examination, some samples will be collected: the natural fluid that comes from the gums and the bacteria that are present there will be collected by inserting a piece of paper and a filter strip in the spaces between teeth and gums; blood samples may also be taken by a phlebotomist to evaluate some inflammatory signs of disease and possible genetic markers (about 5 teaspoons at each visit); and a cheek swab may be taken by gently rubbing a little brush into the inside of the cheeks. Patients also may be asked to spit into a container we provide. Tissues from gums that are usually discarded may also be collected during treatment. When patients return for re-evaluation of their gums, all these samples may be collected again at 3, 6, 12, 18 and 24 months after the initial therapy. After 24 months, only clinical examinations may be performed, up to 3 more visits within the following 3 years.

If the patient does not have gum disease: If gums are healthy and the patient does not need treatment, they will be seen every 6 months for examination and cleanings, then sample collections may also be taken at these visits up to 24 months. These sample collections are done to be studied by genetic tests, which will tell us if there are specific genetic markers (inherited markers) associated with this disease, and also other laboratory testing, which will help the researchers identify how the body responds to bacteria. These markers will also be evaluated in family members (parents, grandparents or siblings), when possible, to check for the likelihood of these members developing this disease.

Regardless of the patient's gum condition, investigators will also evaluate current and past dental x-rays to determine if there were signs of this disease in the past.

Investigators may also take photos of the teeth and gums.

ELIGIBILITY:
Inclusion child/adolescent:

* Male or female, aged 5 to 25
* In good general health as evidenced by medical history
* Diagnosed with localized aggressive periodontitis (LAP), defined by the presence of attachment loss ≥ 2mm and detected bone loss on at least two sites, involving first molars and/or incisors, or
* Periodontally healthy (defined by absence of clinical signs of periodontitis) related or not to LAP participants

Inclusion parent /grandparent:

* Male or female, up to age 90 years
* Parent or grandparent of an enrolled participant with LAP

Exclusion child/adolescent:

* Diagnosed with any systemic diseases or conditions that could influence the progression and/or clinical characteristics of periodontal disease (i.e., immunosuppression, diabetes, neutropenia or blood disorders).
* Patients that have taken antibiotics within the last 3 months* or require antibiotic prophylaxis prior to initial visit.
* Patients that are currently taking medications that could influence the characteristics or response to periodontal treatment (example: immune-suppressive drugs, such as cyclosporine or steroids).
* Smokers (≥10 cigarettes a day for over 6 months)
* Pregnant/lactating women as pregnancy causes gingival changes that could confound study results.
* Any psychiatric conditions that will inhibit participants from proper understanding of study procedures as determined by the PI/clinician investigator.
* Patients may still enroll but will be scheduled for initial visit 3 months later

Exclusion parent/grandparent:

* Patients that have taken antibiotics within the last 3 months* or require antibiotic prophylaxis prior to initial visit.
* Pregnant/lactating women as pregnancy causes gingival changes that could confound study results.
* Any psychiatric conditions that will inhibit participants from proper understanding of study procedures as determined by the PI/clinician investigator.

Ages: 5 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 514 (Actual)
Dates: Start 2006-12 (Actual); Primary Completion 2019-05-29 (Actual); Study Completion 2022-12-02 (Actual)

PRIMARY OUTCOMES:
SNPs and DNA methylation | 24 months
  The investigators are doing analysis of single nucleotide polymorphisms (DNA sequence variation) and methylation (addition of a methyl group) of DNA of specific genes related to inflammation.

SECONDARY OUTCOMES:
Systemic inflammatory levels | 24 months
  The investigators are testing for systemic (plasma levels) and local (gingival fluid levels) markers of inflammation.

CONTACTS AND LOCATIONS:
Overall Officials: Ikramuddin Aukhil, Principal Investigator — University of Florida
Locations (10):
- United States (10):
  - Acorn Dental Clinic, Brooker, Florida
  - Broward College, Fort Lauderdale, Florida
  - Dental Clinical Research Unit, University of Florida, Gainesville, Florida
  - Azalea Dental Clinic, Gainesville, Florida
  - UF Hialeah Dental Clinic, Hialeah, Florida
  - Duval County Department of Health, Jacksonville, Florida
  - UF Naples Pediatric Dental Clinic, Naples, Florida
  - Gadsden County Health Department--Quincy Dental Clinic, Quincy, Florida
  - Leon County Health Department, Tallahassee, Florida
  - University of Kentucky, Lexington, Kentucky

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Albandar JM. Epidemiology and risk factors of periodontal diseases. Dent Clin North Am. 2005 Jul;49(3):517-32, v-vi. doi: 10.1016/j.cden.2005.03.003. PMID 15978239
- [Background] Albandar JM, Tinoco EM. Global epidemiology of periodontal diseases in children and young persons. Periodontol 2000. 2002;29:153-76. doi: 10.1034/j.1600-0757.2002.290108.x. No abstract available. PMID 12102707
- [Background] Albandar JM. Juvenile periodontitis--pattern of progression and relationship to clinical periodontal parameters. Community Dent Oral Epidemiol. 1993 Aug;21(4):185-9. doi: 10.1111/j.1600-0528.1993.tb00753.x. PMID 8370252
- [Background] Sweeney EA, Alcoforado GA, Nyman S, Slots J. Prevalence and microbiology of localized prepubertal periodontitis. Oral Microbiol Immunol. 1987 Jun;2(2):65-70. doi: 10.1111/j.1399-302x.1987.tb00292.x. PMID 10870470
- [Background] Zambon JJ, Christersson LA, Slots J. Actinobacillus actinomycetemcomitans in human periodontal disease. Prevalence in patient groups and distribution of biotypes and serotypes within families. J Periodontol. 1983 Dec;54(12):707-11. doi: 10.1902/jop.1983.54.12.707. PMID 6358452
- [Background] Page RC, Baab DA. A new look at the etiology and pathogenesis of early-onset periodontitis. Cementopathia revisited. J Periodontol. 1985 Dec;56(12):748-51. doi: 10.1902/jop.1985.56.12.748. PMID 3866058
- [Background] Agarwal S, Suzuki JB, Riccelli AE. Role of cytokines in the modulation of neutrophil chemotaxis in localized juvenile periodontitis. J Periodontal Res. 1994 Mar;29(2):127-37. doi: 10.1111/j.1600-0765.1994.tb01101.x. PMID 8158501
- [Background] Christersson LA, Slots J, Rosling BG, Genco RJ. Microbiological and clinical effects of surgical treatment of localized juvenile periodontitis. J Clin Periodontol. 1985 Jul;12(6):465-76. doi: 10.1111/j.1600-051x.1985.tb01382.x. PMID 3894435
- [Result] Shaddox L, Wiedey J, Bimstein E, Magnuson I, Clare-Salzler M, Aukhil I, Wallet SM. Hyper-responsive phenotype in localized aggressive periodontitis. J Dent Res. 2010 Feb;89(2):143-8. doi: 10.1177/0022034509353397. Epub 2009 Dec 30. PMID 20042739
- [Result] Koutouzis T, Haber D, Shaddox L, Aukhil I, Wallet SM. Autoreactivity of serum immunoglobulin to periodontal tissue components: a pilot study. J Periodontol. 2009 Apr;80(4):625-33. doi: 10.1902/jop.2009.080422. PMID 19335083
- [Result] Alfant B, Shaddox LM, Tobler J, Magnusson I, Aukhil I, Walker C. Matrix metalloproteinase levels in children with aggressive periodontitis. J Periodontol. 2008 May;79(5):819-26. doi: 10.1902/jop.2008.070513. PMID 18454660
- [Result] Shaddox LM, Wiedey J, Calderon NL, Magnusson I, Bimstein E, Bidwell JA, Zapert EF, Aukhil I, Wallet SM. Local inflammatory markers and systemic endotoxin in aggressive periodontitis. J Dent Res. 2011 Sep;90(9):1140-4. doi: 10.1177/0022034511413928. Epub 2011 Jul 5. PMID 21730256
- [Result] Shaddox LM, Huang H, Lin T, Hou W, Harrison PL, Aukhil I, Walker CB, Klepac-Ceraj V, Paster BJ. Microbiological characterization in children with aggressive periodontitis. J Dent Res. 2012 Oct;91(10):927-33. doi: 10.1177/0022034512456039. Epub 2012 Aug 3. PMID 22863892
- [Result] Beliveau D, Magnusson I, Bidwell JA, Zapert EF, Aukhil I, Wallet SM, Shaddox LM. Benefits of early systemic antibiotics in localized aggressive periodontitis: a retrospective study. J Clin Periodontol. 2012 Nov;39(11):1075-81. doi: 10.1111/jcpe.12001. Epub 2012 Aug 29. PMID 22931240
- [Result] Goncalves PF, Huang H, McAninley S, Alfant B, Harrison P, Aukhil I, Walker C, Shaddox LM. Periodontal treatment reduces matrix metalloproteinase levels in localized aggressive periodontitis. J Periodontol. 2013 Dec;84(12):1801-8. doi: 10.1902/jop.2013.130002. Epub 2013 Mar 28. PMID 23537121
- [Derived] Branco-de-Almeida LS, Cruz-Almeida Y, Gonzalez-Marrero Y, Kudsi R, de Oliveira ICV, Dolia B, Huang H, Aukhil I, Harrison P, Shaddox LM. Treatment of localized aggressive periodontitis alters local host immunoinflammatory profiles: A long-term evaluation. J Clin Periodontol. 2021 Feb;48(2):237-248. doi: 10.1111/jcpe.13404. Epub 2020 Dec 16. PMID 33205510
- [Derived] Velsko IM, Harrison P, Chalmers N, Barb J, Huang H, Aukhil I, Shaddox L. Grade C molar-incisor pattern periodontitis subgingival microbial profile before and after treatment. J Oral Microbiol. 2020 Sep 13;12(1):1814674. doi: 10.1080/20002297.2020.1814674. PMID 33062199
- [Derived] Harris TH, Wallace MR, Huang H, Li H, Shaddox LM. Associations of P2RX7 Functional Diplotypes with Localized Aggressive Periodontitis. JDR Clin Trans Res. 2019 Oct;4(4):342-351. doi: 10.1177/2380084419863789. Epub 2019 Jul 18. PMID 31319038
- [Derived] Shaddox LM, Mullersman AF, Huang H, Wallet SM, Langaee T, Aukhil I. Epigenetic regulation of inflammation in localized aggressive periodontitis. Clin Epigenetics. 2017 Sep 2;9:94. doi: 10.1186/s13148-017-0385-8. eCollection 2017. PMID 28883894
- [Derived] Branco-de-Almeida LS, Cruz-Almeida Y, Gonzalez-Marrero Y, Huang H, Aukhil I, Harrison P, Wallet SM, Shaddox LM. Local and Plasma Biomarker Profiles in Localized Aggressive Periodontitis. JDR Clin Trans Res. 2017 Jul;2(3):258-268. doi: 10.1177/2380084417701898. Epub 2017 Apr 14. PMID 28879248
- [Derived] Burgess D, Huang H, Harrison P, Aukhil I, Shaddox L. Aggregatibacter actinomycetemcomitans in African Americans with Localized Aggressive Periodontitis. JDR Clin Trans Res. 2017 Jul;2(3):249-257. doi: 10.1177/2380084417695543. Epub 2017 Mar 1. PMID 28879247
- [Derived] Burgess DK, Huang H, Harrison P, Kompotiati T, Aukhil I, Shaddox LM. Non-Surgical Therapy Reduces Presence of JP2 Clone in Localized Aggressive Periodontitis. J Periodontol. 2017 Dec;88(12):1263-1270. doi: 10.1902/jop.2017.170285. Epub 2017 Aug 18. PMID 28820321
- [Derived] Miller KA, Branco-de-Almeida LS, Wolf S, Hovencamp N, Treloar T, Harrison P, Aukhil I, Gong Y, Shaddox LM. Long-term clinical response to treatment and maintenance of localized aggressive periodontitis: a cohort study. J Clin Periodontol. 2017 Feb;44(2):158-168. doi: 10.1111/jcpe.12640. Epub 2016 Dec 27. PMID 27767222
- [Derived] Shaddox LM, Spencer WP, Velsko IM, Al-Kassab H, Huang H, Calderon N, Aukhil I, Wallet SM. Localized aggressive periodontitis immune response to healthy and diseased subgingival plaque. J Clin Periodontol. 2016 Sep;43(9):746-53. doi: 10.1111/jcpe.12560. Epub 2016 Jul 15. PMID 27037664
- [Derived] Allin N, Cruz-Almeida Y, Velsko I, Vovk A, Hovemcamp N, Harrison P, Huang H, Aukhil I, Wallet SM, Shaddox LM. Inflammatory Response Influences Treatment of Localized Aggressive Periodontitis. J Dent Res. 2016 Jun;95(6):635-41. doi: 10.1177/0022034516631973. Epub 2016 Feb 25. PMID 26917438
- [Derived] Merchant SN, Vovk A, Kalash D, Hovencamp N, Aukhil I, Harrison P, Zapert E, Bidwell J, Varnado P, Shaddox LM. Localized aggressive periodontitis treatment response in primary and permanent dentitions. J Periodontol. 2014 Dec;85(12):1722-9. doi: 10.1902/jop.2014.140171. PMID 25186780
- [Derived] Goncalves PF, Klepac-Ceraj V, Huang H, Paster BJ, Aukhil I, Wallet SM, Shaddox LM. Correlation of Aggregatibacter actinomycetemcomitans detection with clinical/immunoinflammatory profile of localized aggressive periodontitis using a 16S rRNA microarray method: a cross-sectional study. PLoS One. 2013 Dec 23;8(12):e85066. doi: 10.1371/journal.pone.0085066. eCollection 2013. PMID 24376864
- [Derived] Shaddox LM, Goncalves PF, Vovk A, Allin N, Huang H, Hou W, Aukhil I, Wallet SM. LPS-induced inflammatory response after therapy of aggressive periodontitis. J Dent Res. 2013 Aug;92(8):702-8. doi: 10.1177/0022034513495242. Epub 2013 Jun 20. PMID 23788609